CLINICAL TRIAL: NCT00523900
Title: Effectiveness of Quaker Complete Nutrition Supplements for Malnourished Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Quaker Oats Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00000428
Record Dates: First submitted 2007-08-31; First posted 2007-09-03 (Estimated); Last update posted 2018-04-03 (Actual); Status verified 2018-03

CONDITIONS: Malnutrition
Keywords: malnutrition; underweight; low body weight; BMI under 19; under nourished; malnourished
MeSH Terms: conditions — Malnutrition; Thinness

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Experimental (Experimental): Malnourished adults who will be given a dietary supplement.
  Interventions: Dietary Supplement: Quaker Complete Nutrition Supplements

INTERVENTIONS:
Dietary Supplement: Quaker Complete Nutrition Supplements — 3-6 250ml cans of Quaker Complete Nutrition Supplements per day

SUMMARY:
Intervention study in malnourished adults to assess whether a nutritional supplement given for 8 weeks in addition to the subject's usual diet improves body weight, body composition, biochemical and immune parameters.

DETAILED DESCRIPTION:
Criteria to be included in this study include:

BMI (Body Mass Index) under 19 Free of cancer, HIV/AIDS, bulimia/anorexia and any malabsorption disorders

Description:

We are studying whether adding nutritional shakes will help participants gain weight and improve their health and immunity. This study lasts about 8 weeks and has a total of 7 visits.

ELIGIBILITY:
Inclusion Criteria:

* BMI (Body Mass Index) under 19
* Adult

Exclusion Criteria:

* HIV/AIDS
* Cancer
* malabsorption disorder

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2007-08; Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
To assess weight-gain efficacy following 8 weeks of dietary supplementation among malnourished adults. | 8 weeks

SECONDARY OUTCOMES:
To compare biochemical and immune markers before and following 8 weeks of treatment with dietary supplements. | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Cheskin, M.D, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins School of Public Health 615 N. Wolfe St Room: E2537, Baltimore, Maryland, United States